CLINICAL TRIAL: NCT07005479
Title: A Prospective Cohort Study on Long-Term Outcomes in Patients With Systemic Lupus Erythematosus at Peking University People's Hospital
Brief Title: Long-Term Outcomes in SLE at Peking University People's Hospital
Acronym: LOTUS
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, He Jing, The Chief of the Rheumatology Department at Peking University People's Hospital, Peking University People's Hospital
Other Study IDs: SLE-PKUPHS
Record Dates: First submitted 2025-05-20; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; LLDAS; survival
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to prospectively follow patients diagnosed with Systemic Lupus Erythematosus (SLE) at Peking University People's Hospital, assessing long-term outcomes such as disease activity, organ involvement, survival, and quality of life. Findings will support individualized patient management and contribute to understanding disease progression in the Chinese population.

DETAILED DESCRIPTION:
This single-center, prospective observational cohort study aims to evaluate the long-term clinical outcomes of patients diagnosed with SLE at Peking University People's Hospital. SLE is a chronic, heterogeneous autoimmune disease that can lead to cumulative organ damage, impaired quality of life, and premature mortality. Although disease control has improved with the advent of immunosuppressive therapies, predicting long-term outcomes remains a challenge.

The study will enroll adult SLE patients and follow them for a period of up to 10 years. Data will be collected at regular intervals, including clinical assessments, laboratory findings, treatment history, and patient-reported outcomes. A particular focus will be placed on measuring disease activity using validated indices such as the SLE Disease Activity Index (SLEDAI) and on evaluating the achievement and maintenance of Lupus Low Disease Activity State (LLDAS).

LLDAS is a validated treat-to-target goal associated with reduced damage accrual and improved prognosis. It will be assessed at each follow-up visit based on established criteria, including low disease activity (SLEDAI-2K ≤4 with no major organ activity), no new disease activity, low-dose glucocorticoid use (prednisone ≤7.5 mg/day or equivalent), and stable standard immunosuppressants. The frequency, duration, and determinants of achieving and sustaining LLDAS over time will be analyzed as a key outcome, alongside major organ involvement, flare rates, survival, and quality of life.

This study will provide real-world data on long-term disease trajectories in a Chinese tertiary hospital population and offer insights into predictors of favorable outcomes, guiding personalized disease management strategies and supporting the implementation of treat-to-target approaches in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* All patients must meet at least one of the following classification criteria for Systemic Lupus Erythematosus (SLE):

The 1997 American College of Rheumatology (ACR) Revised Classification Criteria; The 2012 Systemic Lupus International Collaborating Clinics (SLICC) Classification Criteria; The 2019 EULAR/ACR Classification Criteria for SLE. All patients must be over the age of 18 and competent to provide written consent.

Exclusion Criteria:

* Patients less than 18 years of age and patients who are unable to consent are excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients must be over the age of 18 and competent to provide written consent.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2030-05-20 (Estimated); Study Completion 2032-05-20 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Achieving and Sustaining Lupus Low Disease Activity State (LLDAS) | Approximately 5-10 years
  LLDAS is defined according to the Asia Pacific Lupus Collaboration (APLC) criteria as meeting all of the following at a study visit:
  SLEDAI-2K ≤4 with no activity in major organ systems (renal, CNS, cardiopulmonary, vasculitis, etc.)
  No new features of lupus disease activity compared to the previous assessment
  Physician Global Assessment (PGA) ≤1 (on a 0-3 scale)
  Prednisone (or equivalent) dose ≤7.5 mg/day
  Use of standard maintenance immunosuppressive drugs only

SECONDARY OUTCOMES:
Organ Damage Accrual Measured by the SLICC/ACR Damage Index (SDI) | Annually over a 10-year follow-up period
  Organ damage will be assessed using the Systemic Lupus International Collaborating Clinics/American College of Rheumatology Damage Index (SDI). SDI ranges from 0 to 47, with higher scores indicating more severe, irreversible organ damage accrued since the onset of SLE. A score of 0 indicates no damage, while each additional point reflects cumulative damage in different organ systems.
Lupus-Related Mortality Rate | Approximately 5-10 years
  Number and proportion of deaths directly attributable to SLE or its complications (e.g., infection, renal failure, cardiovascular events).
Glucocorticoid-Sparing Effect | Assessed at each follow-up visit (up to 10 years)
  Proportion of patients achieving and maintaining prednisone (or equivalent) ≤7.5 mg/day without disease flare. Also evaluating cumulative steroid dose over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, Beijing Municipality, China